CLINICAL TRIAL: NCT01700608
Title: Prospective Observational Study on Plerixafor After Chemotherapy
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Paolo Corradini, Professor, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Other Study IDs: 011012
Record Dates: First submitted 2012-10-01; First posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Lymphoma; Myeloma
MeSH Terms: conditions — Lymphoma; Neoplasms, Plasma Cell | interventions — plerixafor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- plerixafor treated patients: lymphoma and myeloma patients
  Interventions: Drug: plerixafor

INTERVENTIONS:
Drug: plerixafor — plerixafor 240 mcg/kg/day at the hematopoietic recovery after chemotherapy
  Other Names: Mozobil

SUMMARY:
Plerixafor is a new CXCR4 inhibitor that is able to improve peripheral blood stem cell (PBSC) mobilization when combined with granulocyte-colony-stimulating factor (G-CSF). The 'on demand' use of plerixafor at the hematopoietic recovery after chemotherapy + G-CSF may be more efficient and cost-effective, but the timing of administration and criteria for patient selection are still under investigation. We collected the data of lymphoma and myeloma patients treated with plerixafor at the hematopoietic recovery after chemotherapy + G-CSF. The decision of adding plerixafor was based on PB CD34+ cells at the time of hematopoietic recovery after chemotherapy in patients at their first or subsequent attempt, according to the attending physician choice. The primary endpoint was the assessment of the rate of patients who were able to collect >=2 x 10^6 CD34+/kg.

DETAILED DESCRIPTION:
Plerixafor is a new CXCR4 inhibitor that is able to improve peripheral blood stem cell (PBSC) mobilization when combined with granulocyte-colony-stimulating factor (G-CSF). The 'on demand' use of plerixafor at the hematopoietic recovery after chemotherapy + G-CSF may be more efficient and cost-effective, but the timing of administration and criteria for patient selection are still under investigation. We collected the data of lymphoma and myeloma patients treated with plerixafor at the hematopoietic recovery after chemotherapy + G-CSF. The decision of adding plerixafor was based on PB CD34+ cells at the time of hematopoietic recovery after chemotherapy in patients at their first or subsequent attempt, according to the attending physician choice. The primary endpoint was the assessment of the rate of patients who were able to collect >=2 x 10^6 CD34+/kg. Secondary endpoint was the assessment of the rate of patients collecting > 4 x 10^6 CD34+/kg and the median number of apheresis to reach the target.

ELIGIBILITY:
Inclusion Criteria:

* lymphoma and myeloma patients treated with plerixafor at the hematopoietic recovery after chemotherapy and G-CSF

Exclusion Criteria:

* patients treated only with G-CSF and plerixafor without chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lymphoma and myeloma patients treated with plerixafor at the hematopoietic recovery after chemotherapy and G-CSF
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2008-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Number of patients who were able to collect >= 2 x 10^6 CD34+/kg | From day 1 to day 25 after mobilizing chemotherapy

SECONDARY OUTCOMES:
Number of patients who were able to collect > 4 x 10^6 CD34+/kg. | From day 1 to day 25 after mobilizing chemotherapy

OTHER OUTCOMES:
To determine the median number of apheresis to reach >= 2-4 x 10^6 CD34+/kg | From day 1 to day 25 after mobilizing chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Corradini, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy, Italy